CLINICAL TRIAL: NCT06801678
Title: Refractive Outcomes Utilizing Two SS-OCT Biometers for IOL Power Calculations
Status: Recruiting | Type: Observational
Sponsor: The Eye institute of Utah (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: 12809-ZJZavodni
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Cataract
Keywords: Biometry; IOL Calculations; ARGOS; IOLM700; SS OCT Biometry
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: No interventions will be administered.

SUMMARY:
The purpose of this study is to evaluate and compare the potential refractive outcomes using the Argos 1.5 biometer in the surgical planning for cataract extraction to that obtained from IOLMaster 700. Both devices are used as standard of care in surgical planning optimization for patients undergoing cataract surgery.

DETAILED DESCRIPTION:
Cataract surgery is one of the most performed surgical procedures globally. The goal of the cataract surgeon is to implant an intraocular lens (IOL) with an appropriate IOL power to compensate for the refractive error and leave the patient emmetropic. The accurate measurement of ocular parameters is therefore critical for the effective calculation of IOL power, which directly impacts postoperative visual outcomes. However, accurate IOL power determination is influenced by several factors, including the measurement techniques employed and the specific biometers used in the process.

Optical biometry has become the gold standard for ocular measurements since the introduction of the IOLMaster (Carl Zeiss Meditec AG, Jena, Germany) in 2001. The IOLMaster 700 utilizes SWEPT Source OCT (SS-OCT) with a wavelength of about 1055 nm to generate a 2D OCT cornea-to-retina cross-section scan of the eye. This allows for the computation of all axial biometry measurements, including axial lengths (AL), central corneal thickness (CCT), anterior chamber depths (ACD), and lens thickness (LT).

A relatively newer biometer, Argos 1.5 is also non-invasive and based on SS-OCT technology for IOL power determination with a similar wavelength of 1060 nm ±10nm. However, the IOLMaster 700 uses a traditional axial length computation approach that relies on a single refractive index whiles Argos 1.5 uses a segmented axial length approach based on multiple refractive indices attributed to each ocular component often referred as True AL.

This study aims to evaluate and compare the potential refractive outcomes and biometric measurements of patients undergoing cataract surgery when using Argos 1.5 versus the IOLMaster 700 with the available formulas on each device. By analyzing these biometric measurements, we aim to uncover insights that could enhance our understanding of how different measurement techniques influence postoperative visual outcomes, ultimately contributing to improved patient care.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older (Adult age)
* Assessed to have Cataract Grade 1 and above per LOCS III or Wisconsin Grading scale in at least one eye.
* Able to comprehend and sign the informed consent form.
* Potential postoperative best corrected distance visual acuity (BCDVA) of 0.3 logMAR or better and targeted post-op refraction to be emmetropia, based on the investigator expert medical opinion.

Exclusion Criteria:

* No active ocular infection or inflammation
* Unable to fixate due to nystagmus or other eye movement abnormality (e.g., significant strabismus)
* Contraindicated for pupil dilation (e.g., narrow angles, allergies) per medical judgement of the investigator.
* Any ocular disease and/or condition that, in the investigator's clinical judgment, may put the subject at significant risk, may compromise study result or may interfere significantly with the subject's participation in the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects at least 21 years of age, meeting inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-02-07 (Estimated); Study Completion 2025-02-22 (Estimated)

PRIMARY OUTCOMES:
Differences in predicted refraction | 1 month
  Predicted refraction is defined as the refractive power predicted by the IOL calculation formula. The predicted refraction for planned IOL power when using Argos 1.5 will be compared to IOL Master 700 for available formulae common to both devices (e.g. SRK/T, Barrett Universal II, Holladay I, Holladay II etc.) using forest plots. Data for Barrett TAL [Argos only] will be analysed using descriptive statistics

SECONDARY OUTCOMES:
Differences in the predicted IOL power for emmetropia | 1 month
  The differences in IOL predicted power will be compared using descriptive statistics and forest plots.
  For the second endpoint, we will be comparing the biometry measurements (ACD, CCT, WTW, LT, AL, K readings) from both devices for the same subject eye. The agreement will be quantified using Bland-Altman analysis for each measure for the total subject population.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary J Zavodni, MD, Principal Investigator — The Eye institute of Utah
Locations (1):
- The Eye Institute of Utah, Salt Lake City, Utah, United States